CLINICAL TRIAL: NCT06027320
Title: Risk Education Technology As Individualized Neuroprotection
Brief Title: The Retain Your Brain Health Study (RetainYourBrain.com)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Retain Health, Inc (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20216157; 4R44AG071416 (NIH)
Record Dates: First submitted 2023-08-25; First posted 2023-09-07 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer Disease; Dementia; Healthy Participants; Brain Health
Keywords: Alzheimer's; Prevention; Clinical Trial
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brain Health Education Arm (Experimental): Subjects will receive an Alzheimer's risk assessment, memory testing, and brain health education, in addition to text message communication.
  Interventions: Behavioral: Brain Health Education
- Alzheimer Disease Education Arm (Other): Subjects will receive an Alzheimer's risk assessment, memory testing, and general education about Alzheimer's disease, in addition to text message communication.
  Interventions: Behavioral: Alzheimer Disease Education

INTERVENTIONS:
Behavioral: Brain Health Education — Subjects will receive an Alzheimer's risk assessment, memory testing, and brain health education, in addition to text message communication.
  Arms: Brain Health Education Arm
Behavioral: Alzheimer Disease Education — Subjects will receive an Alzheimer's risk assessment, memory testing, and general education about Alzheimer's disease, in addition to text message communication.
  Arms: Alzheimer Disease Education Arm

SUMMARY:
The goal of this clinical trial is to test a cell phone-based online program that provides Alzheimer's risk assessments and memory tests over a 6-month period. The main question it aims to answer is whether online software can help reduce the risk of Alzheimer's disease (AD) through digital education and tracking.

Participants will visit RetainYourBrain.com to answer questions about their risk factors for AD and take online word recall and card game cognitive tests. Researchers will track progress over time and compare different strategies of Alzheimer's education to see if it is possible to protect brain health, reduce Alzheimer's risk, and improve memory function.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a public health crisis with few effective treatments. Most people are unaware that AD begins in the brain decades before the first symptoms of memory loss begin. That leaves a lot of time for people to learn their individual risk factors for AD and cognitive decline and take memory assessment screening tests in an effort toward the prevention or delay of dementia. To reach a growing at-risk population, mobile health technologies accessible via cell phone can fill an unmet need due to their accessibility and cost-effective delivery of care. Online education and text messaging have proven to be effective methods of reducing risk for a variety of chronic conditions, including cardiovascular disease and diabetes, which are both key drivers of AD risk.

The investigators created a cell phone-based online software application to provide automated, individualized monitoring and education at broad scale. The goal of the software is to function as a digital therapeutic to identify individual risk factors, assess memory and cognitive function over time, and provide education to people with a family history of AD. The system maintains bi-directional communication via text message to verify participant engagement.

Potential participants who visit our study website (www.RetainYourBrain.com) will be directed to answer questions assessing eligibility criteria. Participants who are eligible are asked to electronically sign an informed consent form, complete baseline assessments, and take online word recall and card game cognitive tests. Participants will then be randomized to one of two groups using different strategies for AD risk assessment education. Researchers will track progress over six months and compare different strategies of education to determine if it is possible to protect brain health, reduce Alzheimer's risk, and improve memory function.

ELIGIBILITY:
Inclusion Criteria:

* be at least 53 years of age
* have a family history of Alzheimer's Disease (AD)
* have a compatible phone/device (phone allowing text messages and with internet access, and/or tablet device with the same capabilities)
* a minimum of one of the following risk factors: body mass index (BMI) of < 25 kg/m2, history of pre-diabetes/diabetes, high blood pressure, high cholesterol, smoking, low physical activity, low fish intake (< 3 times per month), high alcohol intake (< 7 servings per week for a women and <14 servings a week for men), diagnosed with mild or moderate depression.

Exclusion Criteria:

* have a diagnosis of dementia due to AD
* other dementia
* women who are currently pregnant or who plan on becoming pregnant in the next 6 months
* BMI <18.5 kg/m2
* consuming >35 alcoholic drinks/week for men or >28 alcoholic drinks/week for women
* severe depression (PHQ-9 score of more than 15)
* current treatment for cancer
* diagnosis of Parkinson's disease, amyotrophic lateral sclerosis, Lewy body dementia, frontotemporal disorders, multiple sclerosis, or other neurodegenerative disease
* current treatment for an eating disorder
* currently prescribed insulin for type I or II diabetes
* inability to give informed consent or complete identity verification
* participating in another AD trial.

Ages: 53 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 992 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Australian National University Alzheimer's Disease Risk Index (ANU-ADRI) | Baseline, 3 months and 6 months.
  The ANU-ADRI is an evidence-based, validated tool aimed at assessing individual exposure to risk factors known to be associated with an increased risk of developing late-life Alzheimer's Disease (AD). The ANU-ADRI provides an individualized assessment and has been used in studies aiming to evaluate methods of reducing AD risk.

SECONDARY OUTCOMES:
Cogstate Brief Battery | Baseline, 3 months and 6 months.
  The Cogstate Brief Battery (CBB) is a short, internet-based, self-administered cognitive test consisting of four tasks that measure the following cognitive domains: attention, processing speed, learning and working memory. The CBB was developed to detect cognitive changes in the pre-symptomatic stages of AD.
  Psychomotor function is measured by speed of performance (mean of the log10 transformed reaction times for correct responses). Attention is measured by speed of performance (mean of the log10 transformed reaction times for correct responses). Visual learning is measured by accuracy of performance (arcsine transformation of the square root of the proportion of correct responses). Working memory is measured as a speed of performance (mean of the log10 transformed reaction times for correct responses); accuracy of performance (arcsine transformation of the square root of the proportion of correct responses).
Fear of Alzheimer's Disease Scale | Baseline, 3 months and 6 months.
  The FADS is a self-report instrument to directly address anticipatory dementia among a general population of older adults. It assesses 3 main topics: general fear of AD, physiological symptoms accompanying FADS, and worrisome attitudes associated with FADS. In this study, only the general fear subscale will be used with lower scores meaning less fear of Alzheimer's Disease (with 17 being the lowest score and 85 the highest.)

OTHER OUTCOMES:
User Satisfaction | 3 months and 6 months.
  A brief questionnaire will be given to understand how satisfied an individual is with the online software application.
Costs or savings associated with using the online software application | 3 months and 6 months.
  A brief questionnaire will be given to determine if there are any costs or savings associated with using the online software application for brain health education.

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Elgammal, MD, Principal Investigator — Retain Health, Inc; Robert Krikorian, PhD, Principal Investigator — University of Cincinnati School of Medicine; Mark McInnis, BA, Principal Investigator — Retain Health, Inc
Locations (1):
- Retain Health, Inc., Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is an essential part of our proposed activities. We intend to make our results available to the scientific community to contribute to knowledge of the field and avoid unintentional duplication of research. Data from this study will be placed in a research database. Proposals for research will be reviewed by the Principal Investigators, and the data will be made available to qualified researchers via a secure portal.
Supporting Information: Study Protocol, SAP
Time Frame: Six-months after publication of full study results.
Access Criteria: Data will be made available to qualified researchers via a secure portal.
URL: http://www.RetainYourBrain.com

REFERENCES:
- See also: RetainYourBrain Page — http://www.RetainYourBrain.com